CLINICAL TRIAL: NCT03453294
Title: Effect of Trans Nasal Humidified Rapid Insufflation Ventilatory Exchange (THRIVE) During Apneic Oxygenation in General Anesthesia on Biomarkers
Brief Title: Effect of THRIVE During Apneic Oxygenation in General Anesthesia on Biomarkers
Acronym: Bio-THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, Senior Consultant, Associate Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Bio-THRIVE
Record Dates: First submitted 2018-01-21; First posted 2018-03-05 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia; Oxygen Toxicity
Keywords: THRIVE
MeSH Terms: interventions — Intubation, Intratracheal; Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apnoeic oxygenation using THRIVE (Experimental): Oxygenation by apnoea oxygenation using THRIVE
  Interventions: Device: Apnoeic oxygenation using THRIVE
- Endotracheal intubation and mechanical ventilation (Active Comparator): Ventilation and oxygenation by an endotracheal tub and mechanical ventilation
  Interventions: Device: Endotracheal intubation and mechanical ventilation

INTERVENTIONS:
Device: Apnoeic oxygenation using THRIVE — Apnoeic oxygenation using THRIVE
  Arms: Apnoeic oxygenation using THRIVE
Device: Endotracheal intubation and mechanical ventilation — Endotracheal intubation and mechanical ventilation
  Arms: Endotracheal intubation and mechanical ventilation

SUMMARY:
Oxygenation with high-flow nasal cannula with 100% oxygen have now been evaluated in a number of studies and the data are convincing. The THRIVE technique is able to oxygenate patients safely and vital parameters has been shown to be stable. But it is of great importance to evaluate this new concept regarding other potential negative physiological aspects such as biological stress response detected by blood-bourne biomarkers before implementing it into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, >18 years old.
2. Laryngeal-surgery where apnea is of benefit for the surgeon (eg. intraoral or laryngeal surgery).
3. Capable of understanding the study information and sign the written consent.

Exclusion Criteria:

1. American Society of Anaesthesiologist severity score >2
2. New York Heart Association score >2
3. Pacemaker or ICD.
4. Body Mass Index >35
5. Pregnancy
6. Manifest cardiac failure or coronary disease
7. Severe gastrointestinal reflux.
8. Neuromuscular disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Oxidative stress | Up to 2 hours after start of intervention
  Biomarkers of oxidative stress such as Thiobarbituric acid reactive substances, Advanced Oxidation Protein Products,Reactive oxygen species and total antioxidant capacity in blood samples

SECONDARY OUTCOMES:
Biomarkers of neuronal injury | Up to 2 hours after start of intervention
  Biomarkers of neuronal injury and stress in blood such as S100 and Nuclear Serum Enolase
Biomarkers of cardiac damage | Up to 2 hours after start of intervention
  Biomarkers of cardiac damage in blood such as troponin and ProBNP
Biomarkers of kidney injury | Up to 2 hours after start of intervention
  Biomarkers of kidney injury in blood such as creatinine
Markers of RNA damage | Up to 2 hours after start of intervention
  Markers of RNA damage in blood
Inflammatory response | Up to 2 hours after start of intervention
  Biomarkers of Inflammatory response in blood such as cytokines and interleukins

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided